CLINICAL TRIAL: NCT03075709
Title: The Development, Implementation and Evaluation of Clinical Pathways for Chronic Obstructive Pulmonary Disease (COPD) in Saskatchewan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Saskatchewan (Other)
Collaborators: Lung Association of Saskatchewan (Unknown); Novartis (Industry)
Responsible Party: Principal Investigator, Thomas Rotter, Research Chair in Health Quality Improvement Science, University of Saskatchewan
Other Study IDs: BIO-15-286
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Clinical Pathway; CPW; Chronic Obstructive Pulmonary Disease; COPD; Protocol; Adherence; Readmission; Length of Stay; Cost
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Critical Pathways

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Experimental - CPW (Urban): We are working with Regina Qu'Appelle Health Region (RQHR), a primarily urban health region, to develop and implement a clinical pathway (CPW). The CPW will improve care through the following steps: standardizing diagnostic, coordinating and unifying common components of chronic disease care, coordinating the provision of education and reconditioning programs, and ensuring disease specific care utilizes and delivers evidence-informed practices.
  Interventions: Other: Clinical Pathway (CPW)
- Experimental - CPW (Rural): Following implementation in RQHR a rural health region will be chosen as an intervention site for a second CPW. The CPW will improve care through the following steps: standardizing diagnostic, coordinating and unifying common components of chronic disease care, coordinating the provision of education and reconditioning programs, and ensuring disease specific care utilizes and delivers evidence-informed practices.
  Interventions: Other: Clinical Pathway (CPW)
- Control - Standard Care (Urban): Saskatoon Health Region (SHR) will act as the urban control site. No attempts will made to alter care in SHR and therefore patients will continue to receive the current standard of care.
- Control - Standard Care (Rural): Following implementation in RQHR a rural health region will be chosen to act as the rural control site. No attempts will made to alter care in this health region and therefore patients will continue to receive the current standard of care.

INTERVENTIONS:
Other: Clinical Pathway (CPW) — CPWs bring the available evidence to a range of healthcare professionals by adapting guidelines to a local context and detailing the essential steps in the assessment and care of patients.
  Groups: Experimental - CPW (Rural); Experimental - CPW (Urban)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) has substantial economic and human costs. To minimize these costs high quality guidelines have been developed. However, development of guidelines alone rarely results in changes to practice. One method of integrating guidelines into professional practice is the use of clinical pathways (CPWs).

The investigators are working with local stakeholders to develop CPWs for COPD with the aims of improving quality of care and guideline adherence while reducing healthcare utilization. The CPWs will utilize several steps including: standardizing diagnostic training, implementing and unifying common components of chronic disease care, coordinating the provision of education and reconditioning programs, and ensuring disease specific care utilizes and delivers evidence-informed practices. In addition, the investigators have worked to identify evidence-informed strategies for the implementation of the CPWs. Efforts are underway to tailor these implementation strategies for the local context.

The investigators will conduct a three-year quantitative health services research project using an interrupted time series (ITS) design in the form of a multiple baseline approach with control groups. The CPW will be implemented in two Saskatchewan health regions (experimental groups) and two health regions will act as controls (control groups). The experimental and control groups will each contain one urban and one rural health region.

This project is expected to improve quality of life and reduce healthcare utilization. The project will also provide evidence on the effects of CPWs in both urban and rural settings. If the pathways are found effective the investigators will work with all stakeholders to implement similar CPWs for the remaining health regions in the province.

ELIGIBILITY:
Inclusion Criteria:

* All individuals with diagnosed chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The intervention will be implemented at the health region level and will therefore include all individuals diagnosed with chronic obstructive pulmonary disease (COPD) residing within a control or intervention health region.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Care | 36 months
  Operationalized as hospital readmission rates and and emergency department (ED) presentation rates

SECONDARY OUTCOMES:
Healthcare Utilization | 36 months
  Operationalized as hospital admission rates and hospital length of stay
Guideline Adherence | 36 months
  Operationalized as scheduled primary care provider and specialist visits

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Qu'Appelle Health Region, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rotter T, Plishka C, Hansia MR, Goodridge D, Penz E, Kinsman L, Lawal A, O'Quinn S, Buchan N, Comfort P, Patel P, Anderson S, Winkel T, Lang RL, Marciniuk DD. The development, implementation and evaluation of clinical pathways for chronic obstructive pulmonary disease (COPD) in Saskatchewan: protocol for an interrupted times series evaluation. BMC Health Serv Res. 2017 Nov 28;17(1):782. doi: 10.1186/s12913-017-2750-x. PMID 29183318